CLINICAL TRIAL: NCT02021422
Title: A Pilot, Prospective, Non-randomized Evaluation of the Safety of Anakinra Plus Standard Chemotherapy Regimens in Metastatic Pancreatic Ductal Adenocarcinoma Patients
Brief Title: A Pilot, Prospective, Non-randomized Evaluation of the Safety of Anakinra Plus Standard Chemotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 013-018
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Pancreas Cancer
Keywords: metastatic pancreatic ductal adenocarcinoma (PDAC); pancreatic cancer; pancreas cancer; pancreatic adenocarcinoma; metastatic pancreas cancer; metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Interleukin 1 Receptor Antagonist Protein; Oxaliplatin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anakinra with Modified Folfirinox (Other): 8-weeks of anakinra and modified FOLFIRINOX regimen (refer to Appendix 9 for regimen) as follows
  Kineret (anakinra) Dosage Route Administration 100 mg SC Every Other Day
  Modified FOLFIRINOX Drug Dose Administration Oxaliplatin 85 mg/m2 2-4 hours Irinotecan 180 mg/m2 90 minutes fluorouracil 2400 mg/m2 48 hours
  Interventions: Drug: anakinra; Drug: Oxaliplatin; Drug: Irinotecan; Drug: fluorouracil

INTERVENTIONS:
Drug: anakinra — Dosage Route Administration 100 mg SC Every Other Day
  Other Names: Kineret
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 2-4 hours
Drug: Irinotecan — Irinotecan 180 mg/m2 90 minutes
  Other Names: Camptosar
Drug: fluorouracil — fluorouracil 2400 mg/m2 48 hours
  Other Names: 5 FU

SUMMARY:
The study's overall objectives are to evaluate the safety of anakinra in combination with standard chemotherapy regimens in patients with pancreatic ductal adenocarinoma, as well as to collect preliminary immune modulation and clinical activity information, overall survival, and serious adverse events related to the study drug.

DETAILED DESCRIPTION:
Kineret (anakinra) is a FDA-approved drug indicated for rheumatoid arthritis. Anakinra is a recombinant, nonglycosylated form of the human interleukin-1 receptor antagonist (IL-1Ra). Anakinra blocks the biologic activity of IL -1 by competitively inhibiting IL-1 binding to the interleukin-1 type I receptor (IL-1RI), which is expressed in a wide variety of tissues and organs. IL-1 production is induced in response to inflammatory stimuli and mediates various physiologic effects including inflammatory and immunological responses.

This is a pilot, prospective, non-randomized, consecutive enrollment study that will enroll up to 12 subjects who meet the study defined inclusion and exclusion criteria.

Subjects will undergo standard of care chemotherapy treatment/regimens (i.e., modified FOLFIRINOX). Subjects will be dispensed a 2 weeks supply of anakinra the day they begin chemotherapy. They will be instructed to begin self-administering the anakinra (study drug) injections the day after their first dose of chemotherapy.

They will have a blood sample collected at baseline and 6 months follow up. If they have surgery for their disease, they may have a tissue sample collected for later analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Male or non-pregnant and non-lactating female
* Confirmed metastatic/inoperable metastatic pancreas cancer and/or Histologically/cytologically confirmed metastatic adenocarcinoma of pancreas
* Patients' blood counts and blood chemistry levels at baseline must be not clinically significant (NCS) as determined by the enrolling investigator.
* Patient has Eastern Cooperative Oncology Group( ECOG ) Performance Status 0 to 2 (refer to Appendix 5):
* Signed study consent form

Exclusion Criteria:

* <18 years of age
* Pregnant or lactating female
* Patient has islet cell neoplasms
* Active secondary malignancies (2nd cancer not treated/present)
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Known infection with hepatitis B, hepatitis C, or cirrhosis
* Major surgery or vascular device placement (excluding ports for IV medication/chemotherapy) within 2 weeks prior to Day 1 of treatment in study
* History of allergy or hypersensitivity to the study drugs
* Patient is enrolled in any concurrent-outside (outside Baylor University Medical Center or Texas Oncology) clinical protocol or investigational trial
* Significant cardiac disease as defined as New York Heart Association (NYHA) classification III or IV, uncontrolled CHF, or prior MI last 6-months
* Any prior gastrointestinal (GI) disease or history of prior pelvic or abdominal radiation which in the opinion of the investigator may place the patient at increased risk
* Peripheral sensory neuropathy ≥ to grade 2 at baseline
* Significant co-morbidities deemed by investigator as unsuitable for participation/enrollment
* Study consent form not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The Number of Participants with SAEs and AEs. | 6 months
  Test the safety of Anakinra in combination with standard chemotherapy in patients with metastatic pancreatic ductal adenocarcinoma (PDAC) as evidenced by the Number of Participants with serious adverse events (SAEs) and adverse events (AEs).

SECONDARY OUTCOMES:
Overall Survival | 6 months
  Overall Survival (OS) rate as defined by the percentage of people who are alive for a certain period of time after diagnosis
Adverse events associated with injection site reactions and the incidence of infections | 6 Months
  Adverse events associated with injection site reactions and the incidence of infections
Data Collection: tumor measurements by CT scans | 6 months
  Data Collection: tumor measurements by CT scans
Gather preliminary information on the immune modulation and clinical activity of this therapy | 6 month
  * Blood transcriptional profiling
  * Composition of white blood cells
  * Assessment of PDAC antigen--specific T cell repertoire in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Becerra, MD, Principal Investigator — Baylor Sammons Cancer Center
Locations (1):
- Baylor Sammons Cancer Center, Dallas, Texas, United States

REFERENCES:
- [Background] Allantaz F, Chaussabel D, Stichweh D, Bennett L, Allman W, Mejias A, Ardura M, Chung W, Smith E, Wise C, Palucka K, Ramilo O, Punaro M, Banchereau J, Pascual V. Blood leukocyte microarrays to diagnose systemic onset juvenile idiopathic arthritis and follow the response to IL-1 blockade. J Exp Med. 2007 Sep 3;204(9):2131-44. doi: 10.1084/jem.20070070. Epub 2007 Aug 27. PMID 17724127
- [Background] Aspord C, Pedroza-Gonzalez A, Gallegos M, Tindle S, Burton EC, Su D, Marches F, Banchereau J, Palucka AK. Breast cancer instructs dendritic cells to prime interleukin 13-secreting CD4+ T cells that facilitate tumor development. J Exp Med. 2007 May 14;204(5):1037-47. doi: 10.1084/jem.20061120. Epub 2007 Apr 16. PMID 17438063
- [Background] Beatty GL, Chiorean EG, Fishman MP, Saboury B, Teitelbaum UR, Sun W, Huhn RD, Song W, Li D, Sharp LL, Torigian DA, O'Dwyer PJ, Vonderheide RH. CD40 agonists alter tumor stroma and show efficacy against pancreatic carcinoma in mice and humans. Science. 2011 Mar 25;331(6024):1612-6. doi: 10.1126/science.1198443. PMID 21436454
- [Background] Bennett L, Palucka AK, Arce E, Cantrell V, Borvak J, Banchereau J, Pascual V. Interferon and granulopoiesis signatures in systemic lupus erythematosus blood. J Exp Med. 2003 Mar 17;197(6):711-23. doi: 10.1084/jem.20021553. PMID 12642603
- [Background] Chaussabel D, Quinn C, Shen J, Patel P, Glaser C, Baldwin N, Stichweh D, Blankenship D, Li L, Munagala I, Bennett L, Allantaz F, Mejias A, Ardura M, Kaizer E, Monnet L, Allman W, Randall H, Johnson D, Lanier A, Punaro M, Wittkowski KM, White P, Fay J, Klintmalm G, Ramilo O, Palucka AK, Banchereau J, Pascual V. A modular analysis framework for blood genomics studies: application to systemic lupus erythematosus. Immunity. 2008 Jul 18;29(1):150-64. doi: 10.1016/j.immuni.2008.05.012. PMID 18631455
- [Background] Coussens LM, Zitvogel L, Palucka AK. Neutralizing tumor-promoting chronic inflammation: a magic bullet? Science. 2013 Jan 18;339(6117):286-91. doi: 10.1126/science.1232227. PMID 23329041
- [Background] De Monte L, Reni M, Tassi E, Clavenna D, Papa I, Recalde H, Braga M, Di Carlo V, Doglioni C, Protti MP. Intratumor T helper type 2 cell infiltrate correlates with cancer-associated fibroblast thymic stromal lymphopoietin production and reduced survival in pancreatic cancer. J Exp Med. 2011 Mar 14;208(3):469-78. doi: 10.1084/jem.20101876. Epub 2011 Feb 21. PMID 21339327
- [Background] Kalos M, Levine BL, Porter DL, Katz S, Grupp SA, Bagg A, June CH. T cells with chimeric antigen receptors have potent antitumor effects and can establish memory in patients with advanced leukemia. Sci Transl Med. 2011 Aug 10;3(95):95ra73. doi: 10.1126/scitranslmed.3002842. PMID 21832238
- [Background] Kuraishy A, Karin M, Grivennikov SI. Tumor promotion via injury- and death-induced inflammation. Immunity. 2011 Oct 28;35(4):467-77. doi: 10.1016/j.immuni.2011.09.006. PMID 22035839
- [Background] La Torre M, Nigri G, Ferrari L, Cosenza G, Ravaioli M, Ramacciato G. Hospital volume, margin status, and long-term survival after pancreaticoduodenectomy for pancreatic adenocarcinoma. Am Surg. 2012 Feb;78(2):225-9. PMID 22369834
- [Background] Laheru D, Jaffee EM. Immunotherapy for pancreatic cancer - science driving clinical progress. Nat Rev Cancer. 2005 Jun;5(6):459-67. doi: 10.1038/nrc1630. PMID 15905855
- [Background] Lee HC, Ziegler SF. Inducible expression of the proallergic cytokine thymic stromal lymphopoietin in airway epithelial cells is controlled by NFkappaB. Proc Natl Acad Sci U S A. 2007 Jan 16;104(3):914-9. doi: 10.1073/pnas.0607305104. Epub 2007 Jan 9. PMID 17213320
- [Background] Maker AV, Katabi N, Qin LX, Klimstra DS, Schattner M, Brennan MF, Jarnagin WR, Allen PJ. Cyst fluid interleukin-1beta (IL1beta) levels predict the risk of carcinoma in intraductal papillary mucinous neoplasms of the pancreas. Clin Cancer Res. 2011 Mar 15;17(6):1502-8. doi: 10.1158/1078-0432.CCR-10-1561. Epub 2011 Jan 25. PMID 21266527
- [Background] Palucka AK, Gatlin J, Blanck JP, Melkus MW, Clayton S, Ueno H, Kraus ET, Cravens P, Bennett L, Padgett-Thomas A, Marches F, Islas-Ohlmayer M, Garcia JV, Banchereau J. Human dendritic cell subsets in NOD/SCID mice engrafted with CD34+ hematopoietic progenitors. Blood. 2003 Nov 1;102(9):3302-10. doi: 10.1182/blood-2003-02-0384. Epub 2003 Jul 17. PMID 12869510
- [Background] Palucka AK, Ueno H, Connolly J, Kerneis-Norvell F, Blanck JP, Johnston DA, Fay J, Banchereau J. Dendritic cells loaded with killed allogeneic melanoma cells can induce objective clinical responses and MART-1 specific CD8+ T-cell immunity. J Immunother. 2006 Sep-Oct;29(5):545-57. doi: 10.1097/01.cji.0000211309.90621.8b. PMID 16971810
- [Background] Palucka K, Banchereau J. Cancer immunotherapy via dendritic cells. Nat Rev Cancer. 2012 Mar 22;12(4):265-77. doi: 10.1038/nrc3258. PMID 22437871
- [Background] Pascual V, Allantaz F, Arce E, Punaro M, Banchereau J. Role of interleukin-1 (IL-1) in the pathogenesis of systemic onset juvenile idiopathic arthritis and clinical response to IL-1 blockade. J Exp Med. 2005 May 2;201(9):1479-86. doi: 10.1084/jem.20050473. Epub 2005 Apr 25. PMID 15851489
- [Background] Pedroza-Gonzalez A, Xu K, Wu TC, Aspord C, Tindle S, Marches F, Gallegos M, Burton EC, Savino D, Hori T, Tanaka Y, Zurawski S, Zurawski G, Bover L, Liu YJ, Banchereau J, Palucka AK. Thymic stromal lymphopoietin fosters human breast tumor growth by promoting type 2 inflammation. J Exp Med. 2011 Mar 14;208(3):479-90. doi: 10.1084/jem.20102131. Epub 2011 Feb 21. PMID 21339324
- [Background] Ramilo O, Allman W, Chung W, Mejias A, Ardura M, Glaser C, Wittkowski KM, Piqueras B, Banchereau J, Palucka AK, Chaussabel D. Gene expression patterns in blood leukocytes discriminate patients with acute infections. Blood. 2007 Mar 1;109(5):2066-77. doi: 10.1182/blood-2006-02-002477. Epub 2006 Nov 14. PMID 17105821
- [Background] Sebens Muerkoster S, Werbing V, Sipos B, Debus MA, Witt M, Grossmann M, Leisner D, Kotteritzsch J, Kappes H, Kloppel G, Altevogt P, Folsch UR, Schafer H. Drug-induced expression of the cellular adhesion molecule L1CAM confers anti-apoptotic protection and chemoresistance in pancreatic ductal adenocarcinoma cells. Oncogene. 2007 Apr 26;26(19):2759-68. doi: 10.1038/sj.onc.1210076. Epub 2006 Nov 6. PMID 17086212
- [Background] Vence L, Palucka AK, Fay JW, Ito T, Liu YJ, Banchereau J, Ueno H. Circulating tumor antigen-specific regulatory T cells in patients with metastatic melanoma. Proc Natl Acad Sci U S A. 2007 Dec 26;104(52):20884-9. doi: 10.1073/pnas.0710557105. Epub 2007 Dec 18. PMID 18093940
- [Background] Yu CI, Gallegos M, Marches F, Zurawski G, Ramilo O, Garcia-Sastre A, Banchereau J, Palucka AK. Broad influenza-specific CD8+ T-cell responses in humanized mice vaccinated with influenza virus vaccines. Blood. 2008 Nov 1;112(9):3671-8. doi: 10.1182/blood-2008-05-157016. Epub 2008 Aug 19. PMID 18713944